CLINICAL TRIAL: NCT00793702
Title: An Open Phase I Clinical Trial on the Safety and Risk of Sensitisation by Escalating Doses and Repeated Injections of the rdESAT-6 + rCFP-10 Skin Test Reagent Following Intradermal Administration to Healthy Adults
Brief Title: Safety and Risk of Sensitisation of the rdESAT-6 + rCFP-10 Skin Test Following Repeated Intradermal Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TESEC-01; EUDRACT No.: 2008-001489-96
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2013-01-21 (Estimated); Status verified 2013-01

CONDITIONS: Tuberculosis
Keywords: tuberculosis; diagnosis; ESAT-6; CFP-10; skin test; Skin test for the diagnosis of tuberculosis infection
MeSH Terms: conditions — Tuberculosis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A (Experimental): two injections 0.01 µg rdESAT-6 + rCFP-10 (6 weeks interval)
  Interventions: Biological: rdESAT-6 + rCFP-10
- B (Experimental): two injections 0.01 µg rdESAT-6 + rCFP-10 (12 weeks interval)
  Interventions: Biological: rdESAT-6 + rCFP-10
- C (Experimental): two injections 0.1 µg rdESAT-6 + rCFP-10 (6 weeks interval)
  Interventions: Biological: rdESAT-6 + rCFP-10
- D (Experimental): two injections 0.1 µg rdESAT-6 + rCFP-10 (12 weeks interval)
  Interventions: Biological: rdESAT-6 + rCFP-10
- E (Experimental): one injection 1.0 µg rdESAT-6 + rCFP-10
  Interventions: Biological: rdESAT-6 + rCFP-10

INTERVENTIONS:
Biological: rdESAT-6 + rCFP-10 — rdESAT-6 + rCFP-10 skin test administered intradermally by the mantoux injection technique

SUMMARY:
The primary objective is to assess the safety of three dose levels (0.01, 0.1 and 1.0 µg) of the rdESAT-6 + rCFP-10 skin test reagent when injected into healthy adults. The secondary objective is to assess the risk of sensitisation of 0.01 and 0.1 µg rdESAT-6 + rCFP-10 when injected twice with time intervals of 6 or 12 weeks to healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed an informed consent
2. Is willing and likely to be able to comply with the trial procedures
3. Is female/male non-black adult ≥ 18 years and ≤ 55 years of age
4. Is healthy according to a medical examination, medical history and laboratory investigations at inclusion
5. Is prepared to grant authorized persons access to their medical records

Exclusion Criteria:

1. Has a history of tuberculosis or has had a known contact to a person with active tuberculosis
2. Has a positive QuantiFERON-TB Gold In Tube test result at inclusion
3. Laboratory parameters outside of normal range judged by principal investigator to be clinically significant and/or abnormal glucose or protein levels in a urine sample at inclusion
4. Has been in treatment with a product which is likely to modify the immune response within 3 months prior to the day of inclusion (e.g., immunoglobulin, systemic corticosteroids, methotrexate, azathioprine, cyclosporine, infliximab or blood products)
5. Has been vaccinated with a live vaccine within 6 months prior to the day of inclusion (e.g., MMR, yellow fever, or oral typhoid vaccines)
6. Has a known congenital or acquired immune deficiency
7. Has a disease affecting the lymphoid organs (e.g., Hodgkin's disease, lymphoma, leukemia, sarcoidosis)
8. Is known to be infected with HIV, HBV or HCV
9. Has a severe ongoing viral or bacterial infection that might affect the cell mediated immune response at inclusion
10. Has a C-reactive protein (CRP) level > 50 mg/L
11. Has severe scarring, burn, rash, eczema, psoriasis, or any other skin disease at or near the injection site(s)
12. Has a condition in which repeated blood drawings pose more than minimal risk for the volunteer, such as haemophilia, other coagulation disorders, or significantly impaired venous access
13. Is actively participating in another clinical trial or has participated in previous clinical trials investigating the rdESAT-6 skin test reagent
14. Is pregnant according to urine pregnancy test at inclusion
15. Is a female not willing to use contraceptives or is breastfeeding
16. Has a condition which in the opinion of the investigator is not suitable for participation in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Local and systemic adverse events with onset after the FIRST (0.01, 0.1 and 1.0 µg) or SECOND (0.01 and 0.1 µg) injection | onset between the first injection and 28 days after the second injection

SECONDARY OUTCOMES:
The diameter of induration at the second injection site measured transversely to the long axis of the forearm | 72 hours after the second injection

CONTACTS AND LOCATIONS:
Overall Officials: Pernille Nyholm Tingskov, Study Director — Statens Serum Institut
Locations (1):
- Rigshospitalet, Epidemiklinikken, Copenhagen, Denmark

REFERENCES:
- [Derived] Bergstedt W, Tingskov PN, Thierry-Carstensen B, Hoff ST, Aggerbeck H, Thomsen VO, Andersen P, Andersen AB. First-in-man open clinical trial of a combined rdESAT-6 and rCFP-10 tuberculosis specific skin test reagent. PLoS One. 2010 Jun 25;5(6):e11277. doi: 10.1371/journal.pone.0011277. PMID 20593018